CLINICAL TRIAL: NCT00898534
Title: Effect of Immediate Hemoglobin A1c on Glycemic Control in Children With Type I Diabetes Mellitus
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Michael Agus, MD, Children's Hospital Boston
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 03-07-121
Record Dates: First submitted 2009-05-08; First posted 2009-05-12 (Estimated); Last update posted 2009-05-12 (Estimated); Status verified 2009-05

CONDITIONS: Type 1 Diabetes Mellitus; Glycemic Control
Keywords: Pediatrics; Hemoglobin A1c; Point of Care testing
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Immediate Feedback (Experimental): Subjects receive point-of-care hemoglobin A1c testing prior to their diabetes clinic visit, with results made available to the provider during the visit.
  Interventions: Device: Bayer DCA2000+ Hemoglobin A1c analyzer
- Conventional Feedback (No Intervention): Subjects receive laboratory hemoglobin A1c testing at the clinic visit, with results made available to the provider several days later.

INTERVENTIONS:
Device: Bayer DCA2000+ Hemoglobin A1c analyzer — Point-of-care hemoglobin A1c measurement of blood obtained by fingerstick
  Arms: Immediate Feedback

SUMMARY:
Immediate feedback of hemoglobin A1c (A1c) results to adults with type 1 and 2 diabetes allows more appropriate care decisions at the clinic visit and may improve glycemic control. The investigators' objective is to determine whether immediate feedback of A1c results to children with type 1 diabetes will improve patient care and glycemic control.

DETAILED DESCRIPTION:
Because glycosylated hemoglobin (A1c) has been shown to reflect average glycemia over several months and has a strong predictive value for diabetes complications, routine quarterly measurements is a standard of care in children and adolescents with Type 1 diabetes mellitus. The A1c value determines whether the patient's glycemic targets have been reached or maintained. The availability of the A1c result at the time the patient is seen (point-of-care testing) has been reported in adults with diabetes to result in increased intensification of therapy and improvement in glycemic control in type 1 and insulin-treated type 2 diabetes and in type 2 diabetes. The A1c may also serve as a check on the accuracy of the patient's glucose meter and the validity of the patient's reported self monitored blood glucose (SMBG) results.

In many clinical settings, A1c is determined in a central laboratory on a blood sample obtained by venipuncture and results usually are available one to two business days after the sample is obtained. If the A1c value is different than predicted from a review of available SMBG data at the visit, the practitioner must contact the family to review the results and, revise any care decisions made during the visit. This system is inefficient and fraught with the potential for less than optimal care relating to delays in the practitioner seeing the result, delays in reaching the subject or parents, and absence of the subject's participation in the phone call updating the care plan. Furthermore, many children dread venipuncture, which is often poorly tolerated and makes clinic visits painful, emotionally traumatic and unpleasant experiences.

Because there are no published data on the utility of point-of-care A1c testing in children and adolescents with diabetes, we designed a prospective randomized controlled trial to determine if subjects who received immediate feedback of A1c results at their clinic visits would have a lower A1c as compared to those who received A1c results after the clinic visit. We intend to determine whether immediate feedback of A1c results will enable the clinicians providing diabetes care to make more adjustments to the subject's management plan at the time of the clinic visit, and whether this will lead to fewer communications with the subject/family between visits. Finally we will assess the relative pain caused by fingerstick blood sampling as compared to venipuncture.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes mellitus diagnosed at least 2 years prior to enrollment in study
* Less than 18 years of age

Exclusion Criteria:

* Cystic fibrosis related diabetes
* Type 2 diabetes
* Any other suspected non-type 1 diabetes (e.g., maturity onset diabetes of the young)

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 234 (Actual)
Dates: Start 2003-11; Primary Completion 2005-09 (Actual); Study Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
Hemoglobin A1c | 1 year after enrollment

SECONDARY OUTCOMES:
Hemoglobin A1c | 3, 6, and 9 months after enrollment
Pain rating of hemoglobin A1c test | 3, 6, 9, and 12 months after enrollment
Change in diabetes management (insulin, diet, exercise, glucose self-monitoring) | 3, 6, 9, and 12 months after enrollment
Episodes of severe hypoglycemia | 3, 6, 9, and 12 months after enrollment
Hospital admissions for diabetes related event | 3, 6, 9, and 12 months after enrollment
Number of phone and/or email contacts between practitioner and patient | 3, 6, 9, and 12 months after enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Michael SD Agus, MD, Principal Investigator — Boston Children's Hospital
Locations (1):
- Children's Hospital Boston, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Agus MS, Alexander JL, Wolfsdorf JI. Utility of immediate hemoglobin A1c in children with type I diabetes mellitus. Pediatr Diabetes. 2010 Nov;11(7):450-4. doi: 10.1111/j.1399-5448.2009.00635.x. PMID 20070556